CLINICAL TRIAL: NCT04607798
Title: Clinical Evaluation of the Safety and Efficacy of Using Multi-Polar RF and PEMF Technologies for the Treatment of Symptoms Associated With Vulvovaginal Atrophy
Brief Title: Multi-polar RF and PEMF for Treatment of Vulvovaginal Atrophy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Venus Concept (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS0416K
Record Dates: First submitted 2020-10-22; First posted 2020-10-29 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Genitourinary Syndrome of Menopause; Vulvovaginal Atrophy; Menopause
Keywords: Genitourinary Syndrome of Menopause; Menopause; Multi-polar Radio Frequency; Pulsed Electromagnetic Field; Sexual Dysfunction; Vaginal Laxity
MeSH Terms: conditions — Sexual Dysfunction, Physiological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vulvovaginal treatment (Experimental): Internal vaginal treatment monthly for 3 treatments.
  Interventions: Device: Radiofrequency and pulsed electro-magnetic fields treatment

INTERVENTIONS:
Device: Radiofrequency and pulsed electro-magnetic fields treatment — Radiofrequency and pulsed electro-magnetic fields treatment of the vaginal canal to maintain an internal temperature of approximately 42 C for the proximal thermometer and 45 C for the mid and distal thermometers for 15 minutes.

SUMMARY:
The study evaluates the use of multi-polar radiofrequency (RF) and pulsed electro-magnetic fields (PEMF) energies for the treatment of symptoms related to genitourinary syndrome of menopause (GSM)/vulvovaginal atrophy (VVA). All subjects will receive a total of three internal treatments at four week intervals. Subjects will be followed up at one and four months after treatment is complete.

DETAILED DESCRIPTION:
Largely observed in the post-menopausal population, a significant subset of pre-menopausal and peri-menopausal women are also affected by symptoms associated with GSM, the etiology being similar in that there is an interruption in normal estrogen production resulting in a hypoestrogenic state. Symptoms related to GSM include vaginal dryness, decreased lubrication, decreased vaginal elasticity, irritation and discomfort of the vaginal and vulvar tissues in general that can affect sexual health. Traditional treatments, such as hormone replacement therapy (HRT), are often the treatment of choice however come with potential risks and many women are not suitable candidates, or have contraindications to its use. Development of new technologies to address these concerns is warranted.

RF energy-based treatment for symptoms of GSM has been used with success to promote elasticity restoration and improve moisture of the vaginal mucosa, and is well established in literature for the treatment of facial and neck laxity, stress urinary incontinence and skin tightening of tissue. Several studies show favorable results with improvement of vaginal laxity and sexual function with RF treatment. The addition of pulsed electromagnetic field (PEMF) energy to multi-polar RF therapy has also been shown to enhance the results of the RF therapy.

RF therapy has already been reported to be successful in treatment of symptoms related to elasticity restoration and improve moisture of the vaginal mucosa. This study will investigate whether adding PEMF to RF therapy is safe and efficacious for the treatment of symptoms related to GSM and sexual health.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy female subjects, ≥19 years of age presenting with symptoms associated with GSM/VVA.
2. Requesting treatment for vulvovaginal tissue for improvement of symptoms associated with GSM/VVA, with a score of ˂26.55 on the FSFI.
3. Sexual activity (vaginal intercourse minimum twice per month) in a monogamous relationship.
4. At least one full-term pregnancy (>36 weeks gestation) with vaginal delivery completed at least one year before study enrollment.

Exclusion Criteria:

1. Pregnant or intending to become pregnant during the course of study.
2. Having any active electrical implant anywhere in the body, such as a pacemaker or an internal defibrillator.
3. Having a permanent implant in the treated area (e.g. intrauterine device)
4. Prior use of collagen, fat injections and/or other methods of skin augmentation (enhancement with injected or implanted material) in the treated area within 4-6 weeks of the initial treatment or during the course of the study.
5. Use of retinoids such as oral Isotretinoin (Accutane®) within 6 months of initial treatment or during the course of the study.
6. Any other surgery in treated area within 12 months of initial treatment or during the course of the study.
7. Open laceration, abrasion, bleeding, infection or inflammation of any sort on or in the area to be treated.
8. Active sexual transmitted disease (STD) (e.g. genital Herpes Simplex, condylomata) or vaginosis.
9. Chronic vulvar pain or vulvar dystrophy.
10. History of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or use of immunosuppressive medications, including corticosteroids, 6 months prior to and during the course of the study.
11. Having any form of active cancer at the time of enrollment and during the course of the study.
12. Significant concurrent illness, such as uncontrolled diabetes i.e. any disease state that in the opinion of the Investigator would interfere with the treatment, or healing process.
13. Participation in a study of another device or drug within 1 month prior to study enrollment or during this study, and as per the Investigator's careful discretion, as long as not contradictory to any of the above criteria.
14. Mentally incompetent or evidence of active substance or alcohol abuse.
15. Having any stage 3-4 cystocele, rectocele, enterocele paravaginal defect or major pelvic organ prolapse beyond the hymenal ring.
16. Unstable dosages of medications such as antihypertensives or psychotropics that are known to affect sexuality.
17. Skin piercing in the treatment area.
18. Tattoos in the treatment area.
19. Prior skin treatment with laser in the treated area within 6 months of the initial treatment or during the course of treatment.
20. Prior ablative resurfacing procedure in the treated area with laser or other devices within 12 months of the initial treatment or during the course of treatment.
21. History of keloid formation or poor wound healing in a previously-injured skin area.
22. History of epidermal or dermal disorders (particularly if involving collagen or microvascularity).
23. Menstruation less than 7 days prior to treatment.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2017-10-03 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Vaginal Health Index | Six months
  Clinician assessed improvement in five vaginal parameters; (1) vaginal fluid volume, (2) moisture, (3) vaginal epithelial integrity, (4) elasticity and (5) vaginal pH.
  Assessed by the clinician at each visit with baseline comparison made at the one-month and four-month post-treatment assessments.
pH | Six months
  Clinician assessed improvement (reduction) in vaginal pH with baseline comparison made at the one-month and four-month post-treatment assessments.

SECONDARY OUTCOMES:
Female Sexual Function Index (FSFI) | Six months
  Sexual dysfunction criteria (FSFI score ≤26.55) improvement as defined as increased FSFI > 26.55 with treatment; baseline comparison made at the one-month and four-month post-treatment assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Gronski, PhD, Study Director — Venus Concept
Locations (1):
- Cogerent Laser Clinics Group, Kyiv, Ukraine

REFERENCES:
- [Derived] Kolodchenko Y. Nonablative, Noncoagulative Multipolar Radiofrequency and Pulsed Electromagnetic Field Treatment Improves Vaginal Laxity and Sexual Function. Womens Health Rep (New Rochelle). 2021 Jul 27;2(1):285-294. doi: 10.1089/whr.2021.0020. eCollection 2021. PMID 34327510